CLINICAL TRIAL: NCT04017689
Title: THE ASSESSMENT OF THE EFFECTS OF DIFFERENT INFORMATION TECHNIQUES ON PATIENTS ANXIETY LEVELS IN IMPLANT SURGERY
Brief Title: Evaluation of Verbal and Visual Information Techniques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Funda Bastürk, Master student and research assistant in Oral and Maxillofacial surgery, Necmettin Erbakan University
Other Study IDs: NecmettinEU2
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Verbal Information Group: Verbal Information
- Photo Group: Information by photos
- Video Group: Information by video

SUMMARY:
The aim of this study is to evaluate the effects of preoperative and postoperative anxiety levels on patients using oral information, visual information with surgical photographs and visual information via audio-video. To evaluate anxiety levels, dental anxiety scale (DAS), modified dental anxiety scale (MDAS) and state anxiety scale (STAI-S, STAI-T) scales will be used.

DETAILED DESCRIPTION:
After giving written information about the study, an informed consent form will be distributed to patients who want to participate in the study and they will be asked to sign it. Patients who have signed the consent form will be asked to complete the DAS, MDAS, STAI-T and STAI-S questionnaires in the waiting room to assess preoperative anxiety levels.

Verbal, photos and video information used to inform patients. Patients will be randomly divided into 3 groups. A total of 60 patients with 20 patients in each group will be included in the study. Patients in all groups will be operated by the same surgeon. Oral information will be given to the patients in the first group. In the second group, visual information will be given to the patients by showing the photos of the operation process. Patients in group 3 will also be shown a video of an audio implant operation showing the operation process. The operation video of a previously implanted patient will be watched by the attending physician. This video will begin with the physician informing the patient about the implant and continue with anesthesia. Afterward, the video will be terminated by giving information about the implant operation video and the complications that the patient may encounter and the points to be considered after the operation.

A 7-day pain score will be obtained using the Smiley VAS scale to measure postoperative pain levels and patients will be asked to note how many painkillers they use. In addition, blood pressure and pulse measurements will be taken before and after surgery.

A common text was prepared in all groups in order to provide preoperative information in an ideal way. In group 1, information related to this text will be given orally. In the 2nd and 3rd groups, patients will be informed about the same information as well as visuality.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the investigator's clinic for implant surgery

Exclusion Criteria:

* pregnant patients
* patients using psychiatric drugs
* patients with visual problems

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patients between the ages of 18-55, who will receive 1 or 2 implants
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-14 (Estimated)

PRIMARY OUTCOMES:
anxiety scores | before instruct about surgery and after instruct about surgery and postoperative 7th day
  State-Trait Anxiety Inventory (STAI) scale for state anxiety inculude 20 question trait anxiety and 20 question state anxiety.each question has a point value (1 to 5) and higher point indicate worse anxiety
Visual analog scale (VAS) for pain | immediatly postoperative and postoperative 7th day
  scale to find pain amount , pain scores from 0 to 10 will be taken from patients and higher scores indicate worse pain
dental anxiety scores | before instruct about surgery and after instruct about surgery and postoperative 7th day
  Modified Dental Anxiety Scale (MDAS) for dental anxiety include five question, each questions has a point value (1 to 5) and higher point indicate worse anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, Dr, Study Chair — Necmettin Erbakan University/Dentistry Faculty
Locations (1):
- Necmettin Erbakan University Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No